CLINICAL TRIAL: NCT06631404
Title: Renal Arterial Resistive Index as a Noninvasive Biomarker of Disease Activity in Lupus Nephritis Patients
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doaa Rabea Abdelkarim, resident at rheumatology and rehabilitation department, Sohag University
Other Study IDs: Soh-Med-24-09-07MS
Record Dates: First submitted 2024-10-07; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group SLE: Patients with SLE
  Interventions: Diagnostic Test: renal doppler
- group control: matched healthy subjects
  Interventions: Diagnostic Test: renal doppler

INTERVENTIONS:
Diagnostic Test: renal doppler — doppler srudy on renal arteries bilaterally , and detection of RI of renal artery

SUMMARY:
Systemic Lupus Erthymatosous (SLE) is achronic inflammatory multi system auto immue disease characterized by pathogenic auto anti bodies production against nuclear structures (Bolouri et al.,2022), SLE affecting mainly woemn of childbearing age and is chracterized by unpredictable flares and remissions , disease variety varied from mild episode disorder to arpidly progressive life -threatening illness..

LN is diagnosed by either the presence of proteinuria >0.5g/day. active urinary sediment , or an unexplained rise in serum creatinine there fore , identifying new invasive biomarkers of LN severity and outcome is mandatory, Renal Arterial resistive index ( RRI) is anon invasive biomarker that has been studied as apotential indicator of disease activity in LN patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* SLE patients fulfilling the SLE International Collaborating Clinics (SLICC) classification criteria and matched controls.
* Patients cooperative and can answer questions.
* Patients who are able and willing to give written informed consent.

Exclusion Criteria:

* • Individuals with other autoimmune diseases.

  * Diabetes.
  * Hypertension.
  * Heart failure.
  * Hepatic diseases.
  * Chronic renal failure.
  * Renal artery stenosis.
  * Renal vein thrombosis.
  * Intrarenal arteriovenous fistula.
  * Obstructive nephropathy.
  * Urinary tract obstruction that could affect RI of intra renal arteries.
  * Un cooperative patients.
  * Patients not able and willing to give written informed consent.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Aged ≥18 years.
  * SLE patients fulfilling the SLE International Collaborating Clinics (SLICC) classification criteria and matched controls.
  * Patients cooperative and can answer questions.
  * Patients who are able and willing to give written informed consent.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
doppler for renal artery | 1 year
  resistive index of renal artery

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alforaih N, Whittall-Garcia L, Touma Z. A Review of Lupus Nephritis. J Appl Lab Med. 2022 Oct 29;7(6):1450-1467. doi: 10.1093/jalm/jfac036. PMID 35932197
- [Background] Ameer MA, Chaudhry H, Mushtaq J, Khan OS, Babar M, Hashim T, Zeb S, Tariq MA, Patlolla SR, Ali J, Hashim SN, Hashim S. An Overview of Systemic Lupus Erythematosus (SLE) Pathogenesis, Classification, and Management. Cureus. 2022 Oct 15;14(10):e30330. doi: 10.7759/cureus.30330. eCollection 2022 Oct. PMID 36407159
- [Background] Anders HJ, Saxena R, Zhao MH, Parodis I, Salmon JE, Mohan C. Lupus nephritis. Nat Rev Dis Primers. 2020 Jan 23;6(1):7. doi: 10.1038/s41572-019-0141-9. PMID 31974366
- [Background] Anstee QM, Castera L, Loomba R. Impact of non-invasive biomarkers on hepatology practice: Past, present and future. J Hepatol. 2022 Jun;76(6):1362-1378. doi: 10.1016/j.jhep.2022.03.026. PMID 35589256